CLINICAL TRIAL: NCT03624634
Title: A Pilot Study to Assess the Effects of Concussion on Adolescent Rugby Union Players and the Development of a Concussion Passport
Brief Title: Assessment of the Effects of Concussion on Adolescent Rugby Union Players
Status: Completed | Type: Observational
Sponsor: Sports Surgery Clinic, Santry, Dublin (Other)
Responsible Party: Principal Investigator, Dr Neil Welch ASCC, Head of lab services and research, Sports Surgery Clinic, Santry, Dublin
Other Study IDs: SSC-Concussion-001
Record Dates: First submitted 2017-03-15; First posted 2018-08-10 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Concussion, Mild; Concussion, Intermediate; Concussion, Severe
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample retained for analysis for 24 months and the destroyed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
200 adolescent rugby players (aged 15-19) from the Senior Cup Teams of 5 Rugby Playing schools (Members of Irish Schools Rugby) will be invited to enroll for inclusion in the study. The study will collect data on brain health, including computer based skill testing, eye tracking and balance and on task completion, cover existing tests in the established SCAT 3 alongside response to exercise testing and a clinical examination including baseline blood tests known to influence recovery from concussion in a rugby playing population of adolescent schoolboys.

The initial data will be taken before the 2016/2017 season starts. The volume of rugby training and match play will be recorded along with activity monitoring in general. For those subjects who sustain concussion a dedicated clinic will provide all after care including repeat clinical examination and magnetic resonance imaging along with a graduated return to exercise and a compressive rehabilitation programme at Sports Surgery Clinic (SSC). A Consultant Sports Physician will manage the return to play programme with an exercise, cognitive, balance, eye movement and neck strength programme.

DETAILED DESCRIPTION:
Concussion is a traumatic injury to the brain and is a common condition in those athletes who play a contact sport, such as Rugby Union. It is a complex process in which forces are transmitted to the brain and result in temporary impairment of brain function. Governing bodies have done much good work to improve the recognition of concussion and the removal of those players from the field but there still remains much confusion and a lack of data on what measures can be used to help manage the return to school and play after a concussion.

Currently assessment and management of concussion relies heavily on subjective symptom analysis with little in the way of objective measures to help make decisions on diagnosis and safe return to play time frames. There is growing evidence for objective measures of cognition, balance, oculomotor, brain imaging, blood biomarkers and exercise physiology in assisting with concussion diagnosis and management. The importance of the study is to decide on the minimum level of tracking of pre season data to safely enhance the care for rugby playing schoolboys.

Study Methodology

Preseason Baseline assessment (all participants)

All participants will be invited to complete a preseason screening session at SSC comprising:

1. Online questionnaire including past medical history; playing and injury history; sleep, mood, stress, depression, anxiety, QoL assessments; symptom checklist; and predictive and modifying factor analysis.
2. Computerised cognitive assessment: Participants will be screened at baseline using The Axon Sports Baseline Test: a preseason screening test that measures baseline reaction time, learning and memory skills, attention, concentration and problem solving capacity, which can be used in conjunction with The Axon Sports After Injury Test following a suspected concussion.
3. King-Devick Test: An objective method of evaluating visual tracking and saccades (quick, simultaneous movements of both eyes). It involves reading aloud a series of single digit numbers from left to right on three test cards. Participants are asked to read the numbers on each card from left to right as quickly as possible but without making any errors. The sum of the three test card time scores constitutes the summary score for the entire test. The test cards become progressively more difficult to read due to variability of spacing between the numbers. Both errors in reading and speed of reading are included in deriving a score.
4. Vestibulo-ocular Assessment using ICS Impulse Goggles: The goggles are light-weight USB goggles with a disposable face cushion that allow accurate assessment of oculomotor and vestibular function with accuracy by recording eye movement in response to testing stimulus. The participant will be asked to put on the goggles and make sure they are tight but comfortable. They will then be instructed through a series of tests, some of the tests being performed with vision denied. The total testing time will take approximately 5-10 minutes, depending on symptoms onset. The data is collected by the software programme that comes with the ICS Impulse goggles and can be formulated using Excel format and directly uploaded onto the participant's file.

   (I) Benign Paroxysmal Positional Vertigo (BPPV) is a common clinical vestibular dysfunction that can be diagnosed using the head impulse test (vHIT). The test provides quick, clear-cut side of lesion specific assessment of the vestibuloocular reflex response to stimuli in the high-frequency range, the natural range of head movements. It is the only test that can assess all six semicircular canals of the inner ear. ICS Impulse is the world's first vHIT device to combine gold-standard accuracy with unrivaled patient comfort. This test takes 2 minutes to complete unless the patient becomes symptomatic. In this instance, it is appropriate to wait until nystagmus symptoms resolve before moving head position.

   (II) Oculomotor dysfunction can be assessed using the ICS Impluse Goggles which can help to differentiate between a central or peripheral cause. The three common tests look at are: (i) gaze stability to monitor the eye's ability to focus and stabilize by identifying nystagmus that is evoked without stimulus; (ii) VOR tests provide the ability to assess the vestibulo-ocular reflex by identifying the presence or absence of saccadic eye movement in order to simultaneously test for the co-existence of vestibular and cerebellar pathology and thus diagnose vetibuo-cerebellar disease; and (iii) Skew Deviation test provides the ability to diagnose central disorder primarily brainstem by assessing the patient's ocular alignment using a cover-uncover test with the goggles.

   Each test takes approximately 1 minute to complete.
5. Balance assessment: Balance Error Scoring System, as per current SCAT 3 This test will consist of three twenty second tests with different stances." (I) double leg stance (II) Single leg stance (III) Tandem stance

   Each of the 20-second trials is scored by counting the errors or deviations from the proper stance by the participant. The examiner will begin counting errors only after the individual has assumed the proper start position. The modified BESS is calculated by adding one error point for each error during the three 20-second tests. The maximum total number of errors for any single condition is 10. If a participant commits multiple errors simultaneously, only one error is recorded but the participant should quickly return to the testing position and counting should resume once subject is set. Subjects that are unable to maintain the testing procedure for a minimum of five seconds at the start are assigned the highest possible score, ten, for that testing condition.
6. Neck Strength Testing (I) Cervical range of motion will be assessed in three planes of reference (sagittal, frontal and transverse) using the Cervical Range of Motion Instrument (Performance Attainment Associates, Minnesota, USA), which has been validated in various populations. The participant will be seated on a static chair with adjustable height so that the hips, knee and feet are positioned at 90°, and the head placed in the neutral anatomic position. An initial warm-up and familiarisation session practicing all movements to be assessed (flexion, extension, lateral flexion and rotation) will be performed. Upon instruction, the participant will move their head in the test parameter (looking directly ahead) and hold the end of range position to allow the recording of the angle achieved, following which, the individual will return their head to the neutral position. Three separate measures will be made in each direction, the mean of which will be reported.

   (II) Isometric cervical muscle testing is well validated. Maximal voluntary isometric cervical muscle strength in three planes of reference will be assessed with a custom-built device that includes a head harness from Gatherer Systems, a force transducer that is connected to a load cell and bespoke software system. The test will be performed employing a protocol specifically validated in young rugby players, subjecting the neck to manually controlled linear incremental loading to test positional failure in the absence of pain or neurological symptoms (which stops the test). The head is to be held in the neutral anatomic position at all times throughout the test. Peak isometric force will be logged at the point of head movement with loss of test position. Loading will be applied and data will be recorded at 20Hz. Peak isometric force generated by the musculature will be defined as the maximal load recorded during the test procedure. An average of 3 tests will be reported.
7. Accusway Balance assessment: The AMTI Accusway system for balance and postural sway measurement (Advanced Mechanical Technology, Inc., Watertown, Massachusetts) will be used for collecting the data. The Accusway system consists of a portable force platform and SWAYWIN software for data acquisition and analysis. The system measures ground reaction force and moments in 3 orthogonal directions with a sampling frequency of 50 Hz. These provide the COP coordinates, which enables the calculation of the maximum displacement in the anterior-posterior and medial-lateral direction (Max-AP; Max-ML), the root-mean-square amplitude in anterior-posterior and medial-lateral direction from the centroid in x- and y-axis (RMS-AP; RMS-ML), the mean velocity (MV) and the area of the 95th percentile ellipse (AoE).

   The participant will be asked to stand barefooted, double-legged stance on the platform. Because changes in the Base of Support (BOS) have a substantial effect on postural control; the outlines of both feet will be marked on the plastic cover with a permanent marker in order to obtain standardised individual foot positions for the repeated measurements. After leaving the platform, the individual's BOS will be entered in the Accusway Plus system. Maximal BOS width and hip width, measured at the major trochanter femoris, were recorded with an anthropometric caliper (Lafayette Instrument Company, Lafayette, IN).
8. Exercise Challenge Test (ECT) using the University of Buffalo Protocol: The ECT consists of an incremental treadmill exercise test following a standard Balke protocol until symptom exacerbation or voluntary exhaustion. The treadmill speed is set at 3.3mph at 0.0% incline. After 1 minute the grade increases to 2.0% while maintaining the same speed. At the start of the third minute and each minute thereafter, the grade increases by 1%, maintaining the speed at 3.3mph. In addition to frequent heart rate and blood pressure readings and close observation by a therapist, athletes are asked every minute while on the treadmill whether they are experiencing any worsening symptoms. Exercise testing is terminated if symptom exacerbation occurs or the athlete reaches exhaustion (defined by a rate of perceived exertion). Athletes who exercise to voluntary exhaustion without symptom exacerbation are considered ready for RTP. All tests will be performed by medical staff trained in CPR with access to full resuscitation equipment as per SSC protocol.
9. Activity and sleep monitoring (post Concussion Only) - each participant will be given a Fitbit Activity Monitor which uses a three-dimensional accelerometer to sense user movement. The sensor tracks steps taken and combines it with user data to calculate distance walked, calories burned, floors climbed and activity duration and intensity. It also measures sleep quality by tracking periods of restlessness, how long it takes the wearer to fall asleep and how long they are actually asleep. The data collected will be downloaded at each subsequent visit to SSC.
10. Haematology: Blood will be drawn, labelled and prepared for freezing, and only subsequently analysed. This will be performed by experienced venipuncture staff with full PPE and aseptic technique skills. Testing will occur as per SSC Hospital policy. Blood will be stored in a standardized fashion at -80 degrees C for subsequent analysis and novel biomarker discovery programmes. In athletes diagnosed with concussion a detailed profile will be assessed including NFL, NSE, UCH-L1, MBP, S100B, GFAP and Tau protein on the baseline samples. The blood samples will also have genetic analysis performed to look for genes which are thought to influence outcome and recovery from head injury (APO-E). This will be carried out on de-identified samples and will have no long-term implications for the participants. All blood testing will be retrospective and anonymous and will be used for comparison pre and post concussion. Samples will be destroyed 24 months after collection.

Follow Up of Initial Screening All participants will be given a written report on the day of screening for their parents, themselves and their GP's.

A small proportion of asymptomatic individuals will likely be identified with abnormalities on testing. Any abnormal results detected on MRI or other outcome measures will be followed up by the SSC sports medicine team and where necessary, referral to neurologist or neurosurgeon.

A final report summary with de-identified results will be sent on completion of the study to all schools

Post game assessment (all participants) Immediately following a match all participants will be asked to complete an online symptom score and basic wellness questions

Diagnosing concussion The diagnosis of concussion will be made using the Zurich consensus guidelines and the IRFU Guide to Concussion. A medical doctor must make the diagnosis.

Participants will be asked to attend St. Vincent's University Hospital Emergency Department to be assessed by a senior doctor if:

1. No medical doctor is available at a game or training session where a suspected concussion takes place
2. A participant sustains an injury and has a loss of consciousness, focal neurological deficit, vomiting, worsening symptoms of concussion or participant, parent or coach is concerned

Once the diagnosis of concussion has been made and any urgent medical issues have been dealt with then these athletes will enter the post concussion protocol described below.

Participants diagnosed with Concussion

If the participant has been diagnosed with concussion, reports new concussive symptoms or has a cognitive deficit consistent with a concussion, then they will be assessed as follows:

1. Online questionnaire including concussion symptoms scales: As above
2. Computerised cognitive assessment: Participants will complete the Axon Sports After Injury Test which can be compared to the Axon Sports Baseline Test
3. King-Devick Test: As above
4. Vestibulo-ocular assessment using ICS Impulse Goggles: As above
5. Balance assessment: As above
6. Neck strength testing: As above
7. Haematology: As above
8. Activity and sleep monitoring - The data from the Fitbit Activity monitor will be downloaded
9. Exercise Challenge Test: Buffalo Protocol. As above
10. Daily online wellness measurement and symptom profile

Participants will be asked to attend the SSC Concussion clinics where the post injury assessment protocol will be followed by an assessment by the consultant sports & exercise medicine physician and where necessary, referral to a neurologist. Criteria for onward referral to neurology include MRI changes from baseline, symptoms last longer than three weeks, worsening symptoms or worsening neurology.

All participants will be given a written report on the day of assessment for their parents, themselves and their GP's.

Following their assessment, the athletes will be provided with an individualized rehabilitation programme involving return to school advice followed by a graduated return to learn and ultimately return to sport programme. This is the standard accepted current best treatment for concussion and is not considered an intervention.

It is expected that a minimum of two medical assessments by the sports & exercise medicine consultant will be required during the recovery period (the initial assessment and the pre-return to play assessment) and where necessary some of the outcome measures will need to be repeated.

Returning to play Readiness of athletes returning to play is a challenging issue. Informed by the Zurich Consensus Guidelines the Irish Rugby Football Union (IRFU) produced guidelines for the safe return to play of rugby players. For athletes of this age group the guidelines recommend a minimum rest period of 14days post-concussion. Initial emphasis must be on return to learn. Following this, provided all symptoms have subsided, athletes may return to play if their symptoms do not return during a stepwise programme of increasing intensity of physical activity and contact, which includes light aerobic exercise, sport-specific exercise, noncontact training drills and full-contact training. In this age group the minimum time out of rugby before returning to play is 23 days.

Athletes participating in this study will adhere to the IRFU guidelines. The only deviation from these guidelines will be the implementation of the Exercise Challenge Test (Buffalo Protocol). This will be a necessary step to assess changes in performance post concussion. No athlete will return to play before the recommended 23 days.

ELIGIBILITY:
Inclusion Criteria:

1. Playing Rugby Union aged 15-19
2. Be able to understand and cooperate with testing
3. Have parental or guardian consent available

Exclusion Criteria:

1. Unavailable to attend for preseason screening
2. History of neurological or psychiatric disease

Ages: 15 Years to 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescent rugby players (aged 15-19) from the Senior Cup Teams of 5 Rugby Playing schools (Members of Irish Schools Rugby) will be invited to enroll for inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
1) Clinical assessment - assessing change from baseline and between post-concussion visits | 1 Rugby season -2016-2017. All participants will be assessed in preseason (August 2016 - September 2016). Participants who sustain a concussion will have the assessment repeated within 72hours of the concussion and on a weekly basis until fully recovered
  Assessment by physician to determine diagnosis and return to play time frame
2) Questionnaire - assessing change from baseline and between post-concussion visits | 1 Rugby season -2016-2017. All participants will be assessed in preseason (August 2016 - September 2016). Participants who sustain a concussion will have the assessment repeated within 72hours of the concussion and on a weekly basis until fully recovered
  Questionnaire responses will provide qualitative data
3) Computerised cognitive assessment - assessing change from baseline and between post-concussion visits | 1 Rugby season -2016-2017. All participants will be assessed in preseason (August 2016 - September 2016). Participants who sustain a concussion will have the assessment repeated within 72hours of the concussion and on a weekly basis until fully recovered
  Results described as Valid / Invalid
4) King Devick Test - assessing change from baseline and between post-concussion visits | 1 Rugby season -2016-2017. All participants will be assessed in preseason (August 2016 - September 2016). Participants who sustain a concussion will have the assessment repeated within 72hours of the concussion and on a weekly basis until fully recovered
  Score reported in seconds (s)
5) Vestibulo-ocular assessment - assessing change from baseline and between post-concussion visits | 1 Rugby season -2016-2017. All participants will be assessed in preseason (August 2016 - September 2016). Participants who sustain a concussion will have the assessment repeated within 72hours of the concussion and on a weekly basis until fully recovered
  Will provide qualitative data on saccades
6) Balance assessment (BESS) - assessing change from baseline and between post-concussion visits | 1 Rugby season -2016-2017. All participants will be assessed in preseason (August 2016 - September 2016). Participants who sustain a concussion will have the assessment repeated within 72hours of the concussion and on a weekly basis until fully recovered
  BESS scores are presented as numeric values
7) Neck strength - assessing change from baseline and between post-concussion visits | 1 Rugby season -2016-2017. All participants will be assessed in preseason (August 2016 - September 2016). Participants who sustain a concussion will have the assessment repeated within 72hours of the concussion and on a weekly basis until fully recovered
  Results presented in N and N/kg
8) Accusway balance assessment - assessing change from baseline and between post-concussion visits | 1 Rugby season -2016-2017. All participants will be assessed in preseason (August 2016 - September 2016). Participants who sustain a concussion will have the assessment repeated within 72hours of the concussion and on a weekly basis until fully recovered
  Results presented as Change of pressure velocity (mm/s) and sway path length (mm)
9) Exercise Challenge Test - assessing change from baseline and between post-concussion visits | 1 Rugby season -2016-2017. All participants will be assessed in preseason (August 2016 - September 2016). Participants who sustain a concussion will have the assessment repeated within 72hours of the concussion and on a weekly basis until fully recovered
  Scores obtained for heart rate (bpm), RPE and VO2 (ml/kg)
10) Haematology - assessing change from baseline and between post-concussion visits | 1 Rugby season -2016-2017. All participants will be assessed in preseason (August 2016 - September 2016). Participants who sustain a concussion will have the assessment repeated within 72hours of the concussion and on a weekly basis until fully recovered
  Blood analysed for the following biomarkers: NFL, NSE, UCH-L1, MBP, S100B, GFAP and Tau protein
11) Activity monitoring - assessing change from baseline and between post-concussion visits | 1 Rugby season -2016-2017. All participants will be assessed in preseason (August 2016 - September 2016). Participants who sustain a concussion will have the assessment repeated within 72hours of the concussion and on a weekly basis until fully recovered
  FitBit activity monitor will produce scores for steps taken and distance covered (m)

SECONDARY OUTCOMES:
Time to recover from concussion will be recorded | 1 Rugby season -2016-2017. All participants will be assessed in preseason (August 2016 - September 2016). Participants who sustain a concussion will have the assessment repeated within 72hours of the concussion and on a weekly basis until fully recovered
  Results presented in days

CONTACTS AND LOCATIONS:
Overall Officials: Paul McCrory, Study Director — The Florey Institute of Neuroscience and Mental Health
Locations (1):
- Sports Surgery Clinic, Dublin, Leinster, Ireland

REFERENCES:
- [Derived] Cosgrave C, Fuller C, Franklyn-Miller A, Falvey E, Beirne C, Ryan J, McCrory P. Concussion in adolescent rugby union players: comprehensive acute assessment protocol and development of the SSC concussion passport to monitor long-term health. BMJ Open Sport Exerc Med. 2018 Nov 5;4(1):e000455. doi: 10.1136/bmjsem-2018-000455. eCollection 2018. PMID 30498576